CLINICAL TRIAL: NCT06338345
Title: Pharmacokinetics and Modelling of Beta-Lactam in Patients Undergoing Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO)
Brief Title: Pharmacokinetics and Modelling of Beta-Lactam in ECMO-VA Patients
Acronym: KAMELOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC23.0222
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-01

CONDITIONS: Cardiogenic Shock; Post-cardiac Surgery; Cardiac Arrest; Extracorporeal Membrane Oxygenation Complication; Infections
Keywords: VA-ECMO; Infection; Beta-lactam; Pharmacokinetic; Modelling
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piperacillin Tazobactam (Experimental): 75 patients under VA-ECMO receiving a novel administration of Piperacillin Tazobactam.
  Interventions: Diagnostic Test: Therapeutic drug monitoring of beta-lactam
- Cefepime (Experimental): 75 patients under VA-ECMO receiving a novel administration of Cefepime.
  Interventions: Diagnostic Test: Therapeutic drug monitoring of beta-lactam
- Meropenem (Experimental): 75 patients under VA-ECMO receiving a novel administration of Meropenem.
  Interventions: Diagnostic Test: Therapeutic drug monitoring of beta-lactam

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring of beta-lactam — During the 24 first hours after inclusion, 5 blood samples will be collected to mesure plasmatic concentrations of the studied beta-lactam, of creatinin and of albumin

SUMMARY:
The use of antibiotic therapy is common in intensive care units and primarily involves beta-lactams. Its optimal implementation is made difficult by the pharmacokinetic changes inherent in critically ill patients.

Despite the current recommendations from the French Society of Anesthesiology and Intensive Care (SFAR) and the French Society of Pharmacology and Therapeutics (SFPT), there are no recommendations on prescription modalities for patients under veno-arterial extracorporeal membrane oxygenation (VA-ECMO). The use of antibiotic therapy is common in VA-ECMO patients and their pharmacokinetic variability factors are then exacerbated.

We aim to conduct a prospective, multicenter, interventional study designed to identify predictive factors for failure to achieve therapeutic target circulating concentrations of beta-lactams in patients under VA-ECMO treated with one of the studied beta-lactams

DETAILED DESCRIPTION:
The use of antibiotic therapy is common in intensive care units and primarily involves beta-lactams. Its optimal implementation is made difficult by the pharmacokinetic changes inherent in critically ill patients (fluid resuscitation, use of catecholamines, shock state, organ dysfunctions, especially those involved in drug elimination, implementation of extracorporeal circulations...). It has been demonstrated that delayed initiation of appropriate antibiotic therapy in severe infections is an independent predictor of poor prognosis.

The current joint recommendations from the French Society of Anesthesiology and Intensive Care (SFAR) and the French Society of Pharmacology and Therapeutics (SFPT) formulated in 2018 have codified the implementation of beta-lactam antibiotic therapy in critically ill patients, specifying administration modalities, initial dosages, as well as pharmacological therapeutic monitoring methods (plasma monitoring of the administered molecule after 24-48 hours of administration in all patients for whom pharmacokinetic variability is expected) and target plasma concentrations. However, there are no recommendations on prescription modalities for patients under veno-arterial extracorporeal membrane oxygenation (VA-ECMO).

VA-ECMO is a salvage therapy for cardio-pulmonary support via extracorporeal circulation, used in severe cardiac or respiratory failures. The use of antibiotic therapy is common in these patients. Pharmacokinetic variability factors common to intensive care patients are then exacerbated (massive fluid resuscitation, haemodilution by extracorporeal circulation, adsorption of xenobiotics on the exchange membrane and circuit, intensity of organ failures) while the severity of the patient necessitates immediate optimal antibiotic therapy administration.

The literature on antibiotic pharmacokinetics in patients under VA-ECMO is scarce in the adult population. Two exploratory approaches with distinct objectives can be found:

A "fundamental" approach, aiming to define the pharmacokinetic parameters (apparent volume of distribution, elimination half-life...) specific to each molecule within this population and to compare them with those observed in a reference population.

A "clinical" approach, focusing on the frequency of concentrations within the therapeutic range within the studied population (proportion of patients for whom the measured plasma concentration in practice conforms to the targets formulated in the recommendations).

While this second approach seems to correspond more closely to our clinical practice, there are few studies in this area. Bouglé et al. conducted a prospective monocentric study in 2019, including all patients under ECMO-VA receiving antibiotic therapy. The authors described the frequencies of plasma concentrations exceeding the lower limit of the therapeutic range. Thus, within this population of critically ill patients, where the failure to implement optimal antibiotic therapy is likely a factor of poor prognosis, 50 to 90% of patients did not reach the recommended therapeutic targets for the different beta-lactams studied. Moreover, the study considered overdoses as pharmacokinetic successes, a highly debatable point given the complications inherent in beta-lactam overdoses. However, this pilot study did not focus on factors that could predict failure to achieve target concentrations.

We aim to conduct a prospective, multicenter, interventional study designed to identify predictive factors for failure to achieve therapeutic target circulating concentrations of beta-lactams in patients under VA-ECMO treated with one of the studied beta-lactams

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing VA-ECMO
* Patients requiering initiation of a novel antibiotic therapy with one of the studied beta-lactam (Piperacillin-Tazobactam, Cefepime, or Meropenem) while under VA-ECMO
* With an expected survival exceeding 24 hours
* Patient's or their trusted person's consent

Exclusion Criteria:

* Subject under administrative or judicial surveillance
* Non-affiliation to social insurance
* Pregnant or lactating patient
* Antibiotic therapy of interest already initiated before VA-ECMO implantation
* Contraindication to the use of beta-lactam
* Administration modalities of beta-lactam not compliant with current recommendations
* Subject in exclusion period from another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Predictive factors for failure to achieve target plasma concentrations in patients under VA-ECMO treated with Piperacillin-Tazobactam, Cefepime, or Meropenem. | 1 hour after administration
  Plasmatic concentrations during the 24 first hours following the initiation of the antibiotherapy
Predictive factors for failure to achieve target plasma concentrations in patients under VA-ECMO treated with Piperacillin-Tazobactam, Cefepime, or Meropenem. | 3 hour after administration
  Plasmatic concentrations during the 24 first hours following the initiation of the antibiotherapy
Predictive factors for failure to achieve target plasma concentrations in patients under VA-ECMO treated with Piperacillin-Tazobactam, Cefepime, or Meropenem. | 6 hour after administration
  Plasmatic concentrations during the 24 first hours following the initiation of the antibiotherapy
Predictive factors for failure to achieve target plasma concentrations in patients under VA-ECMO treated with Piperacillin-Tazobactam, Cefepime, or Meropenem. | 12 hour after administration
  Plasmatic concentrations during the 24 first hours following the initiation of the antibiotherapy
Predictive factors for failure to achieve target plasma concentrations in patients under VA-ECMO treated with Piperacillin-Tazobactam, Cefepime, or Meropenem. | 24 hour after administration
  Plasmatic concentrations during the 24 first hours following the initiation of the antibiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDRE BEHOUCHE, MD, Principal Investigator — University Hospital, Grenoble
Locations (5):
- France (5):
  - CHU de Clermont Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Dijon-Bourgogne, Dijon
  - Aphp Pitie Salpetriere, Paris
  - CHU ROUEN - Hôpital Charles-Nicolle, Rouen
  - Hôpital Rangueil - CHU Toulouse, Toulouse

REFERENCES:
- [Background] Leone M, Bourgoin A, Cambon S, Dubuc M, Albanese J, Martin C. Empirical antimicrobial therapy of septic shock patients: adequacy and impact on the outcome. Crit Care Med. 2003 Feb;31(2):462-7. doi: 10.1097/01.CCM.0000050298.59549.4A. PMID 12576952
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Blot SI, Pea F, Lipman J. The effect of pathophysiology on pharmacokinetics in the critically ill patient--concepts appraised by the example of antimicrobial agents. Adv Drug Deliv Rev. 2014 Nov 20;77:3-11. doi: 10.1016/j.addr.2014.07.006. Epub 2014 Jul 15. PMID 25038549
- [Background] Roberts JA, Abdul-Aziz MH, Lipman J, Mouton JW, Vinks AA, Felton TW, Hope WW, Farkas A, Neely MN, Schentag JJ, Drusano G, Frey OR, Theuretzbacher U, Kuti JL; International Society of Anti-Infective Pharmacology and the Pharmacokinetics and Pharmacodynamics Study Group of the European Society of Clinical Microbiology and Infectious Diseases. Individualised antibiotic dosing for patients who are critically ill: challenges and potential solutions. Lancet Infect Dis. 2014 Jun;14(6):498-509. doi: 10.1016/S1473-3099(14)70036-2. Epub 2014 Apr 24. PMID 24768475
- [Background] Shekar K, Roberts JA, Welch S, Buscher H, Rudham S, Burrows F, Ghassabian S, Wallis SC, Levkovich B, Pellegrino V, McGuinness S, Parke R, Gilder E, Barnett AG, Walsham J, Mullany DV, Fung YL, Smith MT, Fraser JF. ASAP ECMO: Antibiotic, Sedative and Analgesic Pharmacokinetics during Extracorporeal Membrane Oxygenation: a multi-centre study to optimise drug therapy during ECMO. BMC Anesthesiol. 2012 Nov 28;12:29. doi: 10.1186/1471-2253-12-29. PMID 23190792
- [Background] Bougle A, Dujardin O, Lepere V, Ait Hamou N, Vidal C, Lebreton G, Salem JE, El-Helali N, Petijean G, Amour J. PHARMECMO: Therapeutic drug monitoring and adequacy of current dosing regimens of antibiotics in patients on Extracorporeal Life Support. Anaesth Crit Care Pain Med. 2019 Oct;38(5):493-497. doi: 10.1016/j.accpm.2019.02.015. Epub 2019 Mar 1. PMID 30831307
- [Background] Lamoth F, Buclin T, Pascual A, Vora S, Bolay S, Decosterd LA, Calandra T, Marchetti O. High cefepime plasma concentrations and neurological toxicity in febrile neutropenic patients with mild impairment of renal function. Antimicrob Agents Chemother. 2010 Oct;54(10):4360-7. doi: 10.1128/AAC.01595-08. Epub 2010 Jul 12. PMID 20625153
- [Background] Kuhn D, Metz C, Seiler F, Wehrfritz H, Roth S, Alqudrah M, Becker A, Bracht H, Wagenpfeil S, Hoffmann M, Bals R, Hubner U, Geisel J, Lepper PM, Becker SL. Antibiotic therapeutic drug monitoring in intensive care patients treated with different modalities of extracorporeal membrane oxygenation (ECMO) and renal replacement therapy: a prospective, observational single-center study. Crit Care. 2020 Nov 25;24(1):664. doi: 10.1186/s13054-020-03397-1. PMID 33239110